CLINICAL TRIAL: NCT05507385
Title: A Brief Intervention Targeting Anhedonia in Adolescents: a Feasibility Randomised Controlled Trial
Brief Title: Imagine a Brighter Future: An Intervention to Improve Positive Emotions in Young People
Acronym: IMAGINE-P
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: King's College London (Other)
Collaborators: Mental Health Research UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMAGINE-POSITIVE
Record Dates: First submitted 2022-05-20; First posted 2022-08-19 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-05

CONDITIONS: Depression; Anhedonia
Keywords: Adolescence; Depression; Anhedonia; Mental Imagery
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomised to an intervention group or the control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: IMAGINE-P (Experimental): Experimental intervention: IMAGINE-POSITIVE targeting positive affect (IMAGINE-P):
  The intervention will combine aspects of Memory Specificity Training (MeST), which includes information about the links between memories and emotions, with Positive Prospective Mental Imagery (PPMI).
  Interventions: Behavioral: IMAGINE-POSITIVE
- Control: (Active Comparator): Control intervention: Non-directive supportive therapy (NDST) consists of individual sessions, with an empathetic, emotionally supportive practitioner and provides non-directive problem solving and monitoring. Using NDST will control for factors that may contribute to change, which are not active components e.g. speaking to an empathetic therapist. NDST will follow treatment guidelines.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: IMAGINE-POSITIVE — The intervention will combine aspects of Memory Specificity Training (MeST), which includes information about the links between memories and emotions, with Positive Prospective Mental Imagery (PPMI), to increase vividness and savouring of positive future images, in order to harness positive affect. IMAGINE-PA will follow a treatment manual and delivery will be accompanied by a therapy workbook.
  Arms: Intervention: IMAGINE-P
Behavioral: Control — Non-directive supportive therapy (NDST) consists of individual sessions, with an empathetic, emotionally supportive practitioner and provides non-directive problem solving and monitoring. Using NDST will control for factors that may contribute to change, which are not active components e.g. speaking to an empathetic therapist. NDST will follow treatment guidelines.
  Arms: Control:

SUMMARY:
Depression is a common mental health problem that often begins during adolescence. Onset during adolescence can be disruptive to schoolwork and social relationships and if left untreated can lead to recurrence during adulthood, as well as the development of other mental health problems. Current treatments for depression (for both adults and young people) largely focus on reducing low mood and do not effectively tackle the other hallmark symptom of depression, anhedonia, which is characterised as a loss of enjoyment/ pleasure for previously enjoyed activities. Anhedonia is associated with increased risk of suicidality, so should be an important treatment target. Whilst some adult treatments are beginning to address anhedonia, little research has focussed on young people. It cannot be assumed that adult treatments will work identically in young people, particularly s their brains are still maturing compared to adults. The aim of this study is to complete a randomised feasibility trial, to see if it is possible to run a brief talking therapy for anhedonia in adolescent depression, by targeting one promising cognitive factor known to contribute to low positive affect: positive future mental imagery

DETAILED DESCRIPTION:
The goal of the project is to develop a brief, manualised intervention for adolescent depression that targets anhedonia through harnessing the ability to imagine positive events. This intervention is designed to be delivered in the school environment by practitioners without extensive training. A feasibility randomised controlled trial (RCT) will be conducted by the doctoral student in the proposed project to assess the acceptability of this intervention in schools.

Principal Research Questions:

The primary question is whether a brief, structured intervention to reduce anhedonia symptomatology in depressed adolescents is feasible and acceptable. This trial will inform whether a full-scale efficacy trial is warranted and provide estimates of effect sizes. The trial's primary aims are:

1. To evaluate recruitment and retention for a future efficacy RCT, for example recruitment rates for schools and participants, attrition rates and outcome measure completion.
2. To gather descriptive data on symptom change to inform future estimates of the number of participants required for a fully powered efficacy RCT.

Background:

Depression is a major public health concern, associated with severe and long-lasting impairment. Many cases of depression start in adolescence with adolescent-onsets associated with greater illness burden than adult-onsets. Whilst psychological intervention in adolescence may prevent the persistence of depression into adulthood and its debilitating consequences, these are rarely available. There is also a consistent failure to produce well-replicated efficacious psychological and pharmacological treatments in adolescent depression. In adults, treatment innovation techniques have tried to focus on specific features, such as anhedonia, that are associated with severity and treatment response. Anhedonia, a loss of pleasure or lack of reactivity to pleasurable stimuli, is a hallmark feature of depression. It is associated with brain reward systems and, in youth, predicts illness severity, suicidality and poor treatment response better than other symptoms of depression. Given these findings and that brain reward systems underlying anhedonia are maturing and stabilising in adolescence focussing on the up-regulation of positive emotion during this developmental juncture could be a beneficial therapeutic approach.

Traditionally, psychological interventions for depression target negative affect in the present and/or past. However, potential deficits in processing positive information, in particular positive future-directed cognitions, may be crucial to alleviate anhedonia and produce enhanced treatment response. Mental imagery is suggested to be a powerful tool to promote changes in positive prospective cognitions. In adolescence, this approach could be particularly beneficial as it is a period when future orientation increases and when individuals rely more on imagery for processing and skill acquisition than in adulthood. Although research in this area in adolescent depression is limited, our findings suggest that having more vivid positive future imagery can protect against depressive symptoms in youth following a recent negative life event. Through a National Institute for Health and Care Research (NIHR) funded project, the investigators have developed a novel brief therapy manual and implementation protocol for adolescents using co-design methodology (Research Ethics Sub-Committee ref: HR-15/16-3548; Project ID: 14884). This targets mental imagery in general (rather than positive future mental imagery, in particular) to attenuate depression symptoms. A case series of 9 participants suggests that this intervention is acceptable and may have clinical utility. However, this intervention targets depression generally rather than anhedonia specifically and has only been delivered by an experienced child clinical psychologist. Therefore, the aim of this project is to develop a brief, manualised intervention that targets anhedonia in adolescents with depression, which can be delivered in schools by practitioners without extensive training.

Intervention:

The investigators will adapt our existing therapy manual to create a manualised protocol that more specifically targets positive future imagery to reduce anhedonia. The existing intervention is a four-session programme involving memory specificity training to increase specificity and access to autobiographical memories, imagery re-scripting to reduce distress from negative images and building of positive images. In order to tackle anhedonia more specifically, the investigators will replace negative imagery re-scripting with elements that target up-regulation of positive emotion and expand and elaborate on positive future imagery generation. These changes will also be informed through discussion with other experts and service-user consultants.

Feasibility randomised controlled trial: As this study will assess feasibility and not efficacy, a power calculation to determine sample size is not appropriate. The sample size (n=32, 16 in each arm) was determined with reference to good practice recommendations. The control condition will be 'non-directive supportive therapy', consisting of individual sessions to provide empathy and emotional support, discussion of participant-initiated options for addressing problems and monitoring of depression. The number and frequency of sessions will be matched across groups to control for non-specific factors contributing to change (e.g. passage of time, rapport with an empathic adult). Blind pre/post assessments will be conducted for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14-19
2. Informed consent
3. Willing and able to engage in psychological therapy and complete assessments
4. scoring above clinical cut-off on the MFQ (33 items; clinical cut-off ≥20, and showing high symptoms of anhedonia, as measured by the SHAPS ( 14 items; abnormal level of hedonic tone>2).

Exclusion Criteria:

1. Diagnosis of learning disability (but not difficulty e.g. dyslexia), diagnosis of Autism Spectrum Disorder, or significant head injury, neurological disorder or epilepsy
2. Unable to fluently communicate in spoken English
3. Unable to give informed consent
4. High levels of current risk
5. Currently receiving therapy (including school counselling)
6. Experiencing psychotic symptoms or depressed in the postnatal period (participants with co-morbid physical illness or non-psychotic disorders such as anxiety will not be excluded)

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome - 1: Uptake by schools | Through study completion, an average of 9 months
  A percentage will be calculated for: the number of schools that express interest in the study divided the number of schools that do take part.
Feasibility outcome - 2: Uptake by participants | Through study completion, an average of 9 months
  This will outcome will be assessed at the different stages of participant uptake:
  1. the number of participants that completed the screen questionnaire divided by the number of students who received the screen questionnaire
  2. the number of participants that accepted the invitation to pre-assessment divided by the number of participants that were eligible for pre-assessment from the screen
  3. The number of participants randomised to intervention divided by the number of participants that completed the pre-assessment
  4. The number of participants that completed the post-assessment divided by the number of participants that were randomised to intervention
Feasibility outcome - 3: Intervention completion | Through study completion, an average of 9 months
  The number of participants successfully completing the intervention
Feasibility outcome - 4: Intervention drop-out | Through study completion, an average of 9 months
  The number of participants that drop-out and the reasons for dropping out
Feasibility outcome - 5: Time Period | Through study completion, an average of 9 months
  Time needed to collect and analyse data
Feasibility outcome - 6: Data completeness at pre-assessment | Through study completion, an average of 9 months
  Data completeness for each questionnaire at pre-assessment
Feasibility outcome - 7: Missing Data at pre-assessment | Through study completion, an average of 9 months
  Data missing and reasons for missing data at pre-assessment
Feasibility outcome - 8: Data completeness at post-assessment | Through study completion, an average of 9 months
  Data completeness for each questionnaire at post-assessment
Feasibility outcome - 9: Missing Data at post-assessment | Through study completion, an average of 9 months
  Data missing and reasons for missing data at post-assessment
Feasibility outcome - 10: Data completeness at follow-up assessment | Through study completion, an average of 9 months
  Data completeness for each questionnaire at follow-up assessment
Feasibility outcome - 11: Missing Data at follow-up assessment | Through study completion, an average of 9 months
  Data missing and reasons for missing data at follow-up assessment
Feasibility outcome - 12: Unexpected adverse effects | Through study completion, an average of 9 months
  The number and nature of unexpected adverse effects will be recorded
Acceptability of the intervention - 1: Open questions for qualitative feedback of the programme | Post-intervention (within 2 weeks of post intervention)
  Qualitative questions on the feedback questionnaire:
  1. What did you think of the programme?
  2. Was there anything that made you more likely or less likely to take part in the programme?
  3. How did you find completing the programme at school?
  4. Was there anything about the programme that you really liked?
  5. Was there anything about the training programme that you really didn't like?
  6. What was the most important thing about the programme for you?
  7. Would you recommend this to others who are experiencing difficulties with mood and self-esteem? If so why? Or why not?
  8. Is there anything else you'd like to say about this programme?
Acceptability of the intervention - 2: Satisfaction with the programme | Post-intervention (within 2 weeks of post intervention)
  Participants indicate how satisfied they were with the programme on a 5-point scale; minimum score: 1; maximum score 5. Higher scores indicate better outcome.
Acceptability of the intervention - 3: Feedback on the number of sessions in the programme | Post-intervention (within 2 weeks of post intervention)
  Participants rate what they thought about the number of session on a 5-point scale. 1 = I would have liked 2+ less; 2= I would have liked 1-2 less; 3= I was happy with the number of sessions; 4= I would have liked 1-2 more; 5= I would have liked 2+ more. Minimum score: 1; maximum score 5.
Acceptability of the intervention - 4: Extend the programme has helped | Post-intervention (within 2 weeks of post intervention)
  Participants rate the extent to which the programme helped them on a 5-point scale. Minimum score: 1; maximum score: 5; higher scores indicate better outcome.
Acceptability of the intervention - 5: Recommend the programme to a friend | Post-intervention (within 2 weeks of post intervention)
  Participants rate if they would recommend the programme to a friend on a 5-point scale. 1= no, definitely not; 2= probably not; 3 = unsure; 4 = yes, probably; 5 = yes, definitely. Minimum score: 1; maximum score 5; higher scores indicate better outcome.

SECONDARY OUTCOMES:
Mood and Feelings Questionnaire | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A 33-item measure of low mood in young people rated on a 3-point Likert scale. Minimum score: 0; maximum score: 66; higher scores indicate worse outcome.
Snaith-Hamilton Pleasure Scale | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A measure of anhedonia, consisting of 14 items rated on a 4-point Likert scale. Minimum score: 0; maximum score: 56; higher scores indicate worse outcome.
Positive and Negative Affect Schedule | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A self-report measure of negative and positive affect and consists of 20-items (10 negative items, 10 positive items) rated on a 5-point Likert scale. On each subscale (negative and positive) minimum score: 10; maximum score: 50. Higher scores indicate greater negative affect and greater positive affect.
The Prospective Imagery Task | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A measure of imagery vividness. It has been adapted for use in young people by (Pile et al., 2018). Fourteen scenarios (7 positive and 7 negative) are presented to participants (e.g. "You will achieve something you wanted to"), who are asked to imagine each happening to them and then rate this mental image on a 5-point scale; 'No image at all' (score of 1) to 'Very clear and detailed' (score of 5). Higher scores indicate greater vividness of future imagery.
Autobiographical Memory Task | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A measure of memory specificity. Participants will be given an example of a specific memory and then asked to give a specific memory to ten cue words (five positive; five negative).
Screen for Child Anxiety Related Disorders | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A self-report measure of anxiety, consisting of 41 items rated on a 3-point Likert scale. Minimum score: 0; maximum score: 82; higher scores indicate worse outcome.
Rosenberg Self Esteem Scale | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A 10-item self-report measure of self-worth, rated on a 4-point Likert scale. Minimum score: 0; maximum score: 30; high scores indicate better outcome.
Children's Response Style Questionnaire | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A 25-item self report measure of response styles, rated on a 4-point scale; 'Almost never' (score of 0) to 'Almost always (score of 3). There are with three response style subscales: rumination, distraction and problem solving. Minimum scores on each subscale is 0. Maximum scores for each subscale: rumination: 39, distraction: 21, problem solving: 15. Higher scores indicate a greater tendency to engage in that response style.
Self Compassion Scale | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A 26-item self-report measure of self compassion, rated on a 5-point scale; 'Almost never' (a score of 1) to 'Almost always' (a score of 5). There are 6 subscales of self-compassion: self-kindness, self-judgement, common humanity, isolation, mindfulness and over identification. There is reverse scoring for subscales of self-judgement, isolation and over identification, as these indicate poorer self-compassion. The Self Compassion Scale is scored by computing a total self-compassion score. This total self-compassion score is calculated by first reverse scoring the negative subscales, then taking a mean of each subscale and then taking an average of the 6 subscale means). Self Compassion Scale Norms: 1.0-2.49 = low self-compassion; 2.5-3.5 = moderate self-compassion; 3.51-5.0 = high self-compassion.
Child Revised Impact of Event Scale | Pre-intervention (baseline), post-intervention (within 2 weeks of post intervention), 3 month follow up
  A 13-item measure of post-traumatic stress symptoms in reference to a recent negative event, rated on a 4-point scale; Not at all (score of 0), Rarely (score of 1), Sometimes (score of 3), Often (score of 5). Minimum score: 0; Maximum score: 65. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan for individual participant data

REFERENCES:
- [Background] Zisook S, Lesser I, Stewart JW, Wisniewski SR, Balasubramani GK, Fava M, Gilmer WS, Dresselhaus TR, Thase ME, Nierenberg AA, Trivedi MH, Rush AJ. Effect of age at onset on the course of major depressive disorder. Am J Psychiatry. 2007 Oct;164(10):1539-46. doi: 10.1176/appi.ajp.2007.06101757. PMID 17898345
- [Background] Bridge JA, Birmaher B, Iyengar S, Barbe RP, Brent DA. Placebo response in randomized controlled trials of antidepressants for pediatric major depressive disorder. Am J Psychiatry. 2009 Jan;166(1):42-9. doi: 10.1176/appi.ajp.2008.08020247. Epub 2008 Dec 1. PMID 19047322
- [Background] Gabbay V, Johnson AR, Alonso CM, Evans LK, Babb JS, Klein RG. Anhedonia, but not irritability, is associated with illness severity outcomes in adolescent major depression. J Child Adolesc Psychopharmacol. 2015 Apr;25(3):194-200. doi: 10.1089/cap.2014.0105. Epub 2015 Mar 24. PMID 25802984
- [Background] Pizzagalli DA. Depression, stress, and anhedonia: toward a synthesis and integrated model. Annu Rev Clin Psychol. 2014;10:393-423. doi: 10.1146/annurev-clinpsy-050212-185606. PMID 24471371
- [Background] Giedd JN. The teen brain: insights from neuroimaging. J Adolesc Health. 2008 Apr;42(4):335-43. doi: 10.1016/j.jadohealth.2008.01.007. PMID 18346658
- [Background] Dunn BD. Helping depressed clients reconnect to positive emotion experience: current insights and future directions. Clin Psychol Psychother. 2012 Jul-Aug;19(4):326-40. doi: 10.1002/cpp.1799. Epub 2012 Jun 5. PMID 22674611
- [Background] Holmes EA, Blackwell SE, Burnett Heyes S, Renner F, Raes F. Mental Imagery in Depression: Phenomenology, Potential Mechanisms, and Treatment Implications. Annu Rev Clin Psychol. 2016;12:249-80. doi: 10.1146/annurev-clinpsy-021815-092925. Epub 2016 Jan 15. PMID 26772205
- [Background] Burnett Heyes S, Lau JY, Holmes EA. Mental imagery, emotion and psychopathology across child and adolescent development. Dev Cogn Neurosci. 2013 Jul;5:119-33. doi: 10.1016/j.dcn.2013.02.004. Epub 2013 Mar 5. PMID 23523985
- [Background] Pile V, Lau JYF. Looking forward to the future: Impoverished vividness for positive prospective events characterises low mood in adolescence. J Affect Disord. 2018 Oct 1;238:269-276. doi: 10.1016/j.jad.2018.05.032. Epub 2018 May 30. PMID 29894932
- [Background] Pile V, Smith P, Leamy M, Blackwell SE, Meiser-Stedman R, Stringer D, Ryan EG, Dunn BD, Holmes EA, Lau JYF. A brief early intervention for adolescent depression that targets emotional mental images and memories: protocol for a feasibility randomised controlled trial (IMAGINE trial). Pilot Feasibility Stud. 2018 Jul 4;4:97. doi: 10.1186/s40814-018-0287-3. eCollection 2018. PMID 29997904
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT05507385/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT05507385/ICF_001.pdf